CLINICAL TRIAL: NCT03899389
Title: Plasma TMAO (Trimethylamine N-oxide) as a Predictive Marker in Coronary Disease Patients
Status: Completed | Type: Observational
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Principal Investigator, Robert Olek, Associate Professor, Gdansk University of Physical Education and Sport
Other Study IDs: DSRiK/10/2018
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Coronary Disease
Keywords: trimethylamine-N-oxide
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute Coronary Syndrome (ACS): Patients with STEMI or NSTEMI infarction, who were admitted to the hospital with chest pain.
  Interventions: Diagnostic Test: plasma samples collection
- Stable Angina (SA): Patients with stable angina who were scheduled for conventional coronary angiography.
  Interventions: Diagnostic Test: plasma samples collection
- Control Group (CON): Healthy control group responding by age and gender to examined groups.
  Interventions: Diagnostic Test: plasma samples collection

INTERVENTIONS:
Diagnostic Test: plasma samples collection — Trimethylamine N-oxide (TMAO) concentration will be determined in plasma samples

SUMMARY:
The primary aim of the current research project is to determine whether the TMAO concentration in the blood can serve as a prognostic indicator of myocardial infarction.

The hypothesis is that in patients with recent myocardial infarction, TMAO concentration in blood is higher than in patients undergoing scheduled coronarography.

DETAILED DESCRIPTION:
To the study will be included volunteers - patients with stable angina (SA), who were scheduled for conventional coronary angiography, and patients with acute coronary syndrome (ACS) who were admitted to the hospital with chest pain and undergoing coronography surgery. Blood samples will be taken from volunteers once - before the coronography surgery by qualified medical personnel.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed stable angina (SA) or acute coronary syndrome (ACS) and planned coronography

Exclusion Criteria:

* unconscious patient

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Pomeranian Cardiology Centers in Wejherowo
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Trimethylamine-N-oxidec(TMAO) blood concentration | Immediately before coronography.
  TMAO concentration determined by the ultra-performance liquid-chromatography tandem mass spektrometry (UPLC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olek, PhD, Principal Investigator — University of Physical Education and Sport in Gdansk
Locations (1):
- University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No